CLINICAL TRIAL: NCT05889507
Title: Whole-body Hypothermia Versus Normothermia in Mild Neonatal Encephalopathy: A Multicentre Randomised Controlled Trial
Brief Title: Cooling in Mild Encephalopathy
Acronym: COMET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 326176
Record Dates: First submitted 2023-05-12; First posted 2023-06-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Encephalopathy; Newborn Asphyxia
Keywords: therapeutic hypothermia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Administration of cooling therapy cannot be masked. The 24 (±2) months of age assessments will be performed by a central team of 2 to 3 examiners, masked to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body hypothermia (Experimental): Whole-body hypothermia (33.5±0.5°C) will be initiated within 6 hours of birth and continued for 72 hours using a servo-controlled cooling machine at the nearest available neonatal intensive care unit (cooling centre).
  Interventions: Procedure: Whole body hypothermia; Other: Supportive neonatal intensive care; Diagnostic Test: Follow up assessment at 2 years of age
- Normothermia (Active Comparator): The axillary temperature will be maintained at 37±0.5°C using servo-controlled incubators for the first 80 hours and any hyperthermia will be treated with a standardised protocol.
  Interventions: Procedure: Targeted normothermia; Other: Supportive neonatal intensive care; Diagnostic Test: Follow up assessment at 2 years of age

INTERVENTIONS:
Procedure: Whole body hypothermia — Whole-body hypothermia (33.5±0.5°C) initiated within 6 hours of birth and continued for 72 hours. The rectal temperature will be maintained at 33.5±0.5°C using a servo-controlled cooling machine.
  Arms: Whole body hypothermia
Procedure: Targeted normothermia — The axillary temperature will be maintained at 37±0.5°C for the first 80 hours and any hyperthermia will be treated with a standardised protocol.
  Arms: Normothermia
Other: Supportive neonatal intensive care — Neonatal intensive care monitoring and support including ventilatory and inotropic support as clinically indicated
Diagnostic Test: Follow up assessment at 2 years of age — The assessment will be carried out using the Bayley Scales of Infant and Toddler Development IV. In addition, all infants will have a detailed neurological examination, including Gross Motor Function Classification System (GMFCS) for cerebral palsy, vision, and hearing assessment. Babies who die or who cannot be assessed with the Bayley-IV due to severe disability will be allocated a Cognitive Scale Composite score one point below the basal test score. PARCA-R will be completed by the parents immediately.

SUMMARY:
The goal of this randomised control trial is to establish the safety and efficacy of whole-body hypothermia for babies with mild hypoxic ischaemic encephalopathy, inform national and international guidelines, and establish uniform practice across the NHS.

The main questions it aims to answer are:

1. Does whole-body cooling (33.5±0.5°C) initiated within six hours of birth and continued for 72 hours, improve cognitive development at 24 (±2) months of age after mild neonatal encephalopathy compared with normothermia (37±0.5°C)?
2. Does a prospective trial-based economic evaluation support the provision of cooling therapy for mild encephalopathy in the NHS on cost-effectiveness grounds?

Participants will have the following interventions:

* Randomisation into one of the following groups

  * Whole body hypothermia group
  * Targeted normothermia group
* Bayley Scales of Infant and Toddler Development 4th Edition (Bayley-IV) examination at 24 (±2) months of age.

Researchers will compare the mean Cognitive Composite Scale score from the Bayley IV examination between the two groups.

DETAILED DESCRIPTION:
COMET is a phase III prospective multi-centre open label two-arm randomised controlled trial with an internal pilot and masked outcome assessments. Administration of cooling therapy cannot be masked.

All babies born at or after 36 weeks and requiring prolonged resuscitation at birth (defined as continued resuscitation at 10 minutes after birth or 10-minute Apgar score less than 6) or those with severe birth acidosis (defined as any occurrence of: pH =<7.00 or Base deficit >=16mmol/l in any cord or baby gas sample within 60 minutes of birth) and admitted to the neonatal unit will started on aEEG or EEG as a part of standard clinical care.

Neonatal doctors or advanced nurse practitioners (clinical team) will screen for eligibility using a structured neurological examination performed between 1 to 6 hours after birth.

Once parental consent is obtained, babies will be randomised to whole-body hypothermia or targeted normothermia within 6 hours of birth, using a web-based program. Initial assessment and randomisation (and initiation of whole-body hypothermia or targeted normothermia) will occur at the hospital of birth. The babies in both arms, who are born at a non-cooling centre (LNU or SCBU) will be then transferred to the nearest cooling centre (NICU) within 8 hours of birth for continued care.

Whole-body hypothermia (33.5±0.5°C) will be initiated within 6 hours of birth and continued for 72 hours using a servo-controlled cooling machine at the nearest available neonatal intensive care unit (cooling centre). Passive cooling methods will not be allowed. Whole-body hypothermia to 33.5±0.5°C for 72 hours is the duration and depth of cooling that is standard for babies with moderate or severe HIE in high income countries. To administer this intervention babies will be kept on a cooling mattress or blanket circulating a coolant/water, a rectal temperature probe will be inserted, and overhead radiant warmers will be switched off. The cooling device will be set to hypothermia mode and body temperature will be rapidly reduced to 33.5°C from 37.0°C and maintained within the target range of 33°C to 34°C.

In the Normothermia (Control group), the rectal temperature will be maintained at 37.0±0.5°C for the first 88 hours and any hyperthermia will be treated with a standardised protocol. Four hourly axillary temperature will be recorded during the first 88 hours. Babies in the control group who develop seizures (level 1 or level 2) and progress to moderate HIE between 6 to 24 hours may be treated with whole-body cooling for 72 hours as clinical care, although this is expected to occur in less than 5%.

Conventional MRI using standard 3D T1-weighted and 2D T2-weighted sequences and diffusion weighted imaging will be performed prior to discharge home.

The follow-up assessment will be done when the recruited babies are 24 (±2) months of age. The assessment will be carried out using the Bayley Scales of Infant and Toddler Development IV. It is a validated and standardized scoring system that assesses development in three domains, that is cognition, language, and motor development. In addition, all infants will have a detailed neurological examination, including Gross Motor Function Classification System (GMFCS) for cerebral palsy, vision, and hearing assessment. Babies who die (the mortality rate is expected to be less than 1% in mild HIE) or who cannot be assessed with the Bayley-IV due to severe disability will be allocated a Cognitive Scale Composite score one point below the basal test score (i.e., score of 54). In all infants, PARCA-R (online or face to face) will be completed by the parents immediately prior to the Bayley IV assessments and CBCL (face to face only) after the Bayley IV assessments.

The data will be collected into a paper case report form (CRF) initially and then entered into electronic database at the participating sites. Data will include ante-natal, birth, and neonatal clinical information including gestational age, birth weight, gender, Apgar scores, birth history, delivery room resuscitation to assess the baseline comparability of the groups, core body temperature for assessment of intervention, details of the hospital course, laboratory investigations and MR imaging for safety monitoring, and neurodevelopmental outcomes at 24 (±2) months of age for primary outcome evaluation.

ELIGIBILITY:
Inclusion Criteria:

All babies born at or after 36 weeks of gestation with a birth weight of 1800g or more with birth acidosis or requiring resuscitation at birth will be screened for eligibility.

Parents will be approached for consent if the baby meets all the three (A + B + C) criteria below:

A. Evidence of intra-partum hypoxia-ischemia defined as any of - (i) Apgar score of <6 at 10 minutes after birth; (ii) continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth; (iii) severe birth acidosis defined as any occurrence of pH =<7.00 or a Base deficit >=16mmol/l in any cord or baby gas sample within 60 minutes of birth.

B. Evidence of mild hypoxic ischaemic encephalopathy defined as - two or more abnormal findings in any of the six categories of the modified Sarnat examination (level of consciousness, spontaneous activity, posture, tone, primitive reflexes, and autonomic nervous system) but not meeting the diagnosis of moderate or severe hypoxic ischaemic encephalopathy on a standardised examination performed by a certified examiner between 1 to 6 hours of age.

C. Normal amplitude on aEEG performed for at least 30 minutes between 1 to 6 hours of age. Normal amplitude will be defined as upper margin of the aEEG activity more than 10 microvolts and the lower margin more than 5 microvolts on a single channel aEEG.

Exclusion Criteria:

* Infants who meet the BAPM criteria for whole-body hypothermia
* Infants without encephalopathy defined as less than two abnormalities on structured neurological examination.
* Infants with major congenital or chromosomal anomalies identified prior to randomisation.
* Infants with birthweight <1800g.
* Infants who have already received sedation, muscle relaxation, or anti-convulsants prior to neurological assessment.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 426 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean Cognitive Composite Scale score from the Bayley IV examination | 22 to 26 months
  The Bayley scales of Infant and toddler development IV is a validated and standardised scoring system that assesses development of three domains, that is cognition, language, and motor development. Babies who die or who cannot be assessed with the Bayley IV due to severe disability will be allocated a Cognitive Scale Composite score one point below the basal test score similar to the previous whole-body hypothermia trials.

SECONDARY OUTCOMES:
Neonatal seizures | During neonatal hospitalisation (Expected average of 2 weeks)
  Definite seizures: seizures confirmed on EEG with or without clinical manifestations or Level 2-Probable seizure: clinically assessed focal clonic/ focal tonic seizure or seizures confirmed on aEEG.
Duration of intensive care. | During neonatal hospitalisation (Expected average of 2 weeks)
  Number of days of neonatal intensive care.
Duration of hospital stay. | During neonatal hospitalisation (Expected average of 2 weeks).
  Total number of days of inpatient care in a neonatal unit.
Duration of mechanical ventilation. | During neonatal hospitalisation (Expected average of 2 weeks).
  Number of hours on invasive ventilation through an endotracheal tube.
Duration of inotropic support. | During neonatal hospitalisation (Expected average of 2 weeks).
  Total number of hours on inotropic support.
Number of babies with bloodstream or cerebrospinal fluid positive infection. | During neonatal hospitalisation (Expected average of 2 weeks).
  Isolation of a pathogenic organism from blood or cerebrospinal fluid along with a clinical diagnosis of sepsis, at any time during neonatal hospitalisation.
Number of babies with thrombocytopenia or coagulopathy requiring transfusion of blood products. | During neonatal hospitalisation (Expected average of 2 weeks).
  Prolonged blood coagulation requiring blood products
Opioid use. | During neonatal hospitalisation (Expected average of 2 weeks).
  Total cumulative dose of morphine per kilogram of body weight.
Number of babies exclusively breastfeeding at hospital discharge. | During neonatal hospitalisation (Expected average of 2 weeks).
  Defined as the newborn receiving only breast milk the last feedings before discharge.
Brain injury scores on conventional magnetic resonance imaging | During neonatal hospitalisation (Expected average of 2 weeks).
  Defined as per Rutherford/NICHD staging.
Survival without any neurological impairment. | 22 to 26 months
  Score of >85 in all Bayley-IV domains (motor, language, and cognitive), normal neurological examination with no cerebral palsy (Gross motor function classification system score <1), no hearing or visual impairment (as reported by parents), and no seizure disorder.
Preschool Child Behaviour Checklist (CBCL 1½-5) | 22 to 26 months
  Completed by parents at the 24-month assessment to provide a standardised measure of children's behavioural outcomes on scales that assess internalizing and externalizing behaviour problems and a Total Problems Scale. Mean standardised T-scores on each scale will be compared between groups. The CBCL checklist will be completed after the Bayley IV assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, PhD, Principal Investigator — Imperial College London; Seetha Shankaran, MD, Principal Investigator — Wayne State University
Locations (39):
- Neonatal Unit, Università degli Studi della Campania "Luigi Vanvitelli", Naples, Italy
- United Kingdom (38):
  - William Harvey Hospital, Ashford
  - St Peters Hosptial, Ashford
  - Birmingham Heartlands, Birmingham
  - Royal Bolton Hosptial, Bolton
  - Bradford Royal Infirmary, Bradford
  - Royal Sussex County Hospital, Brighton
  - St Michael's Hospital, Bristol
  - Southmead Hosptial, Bristol
  - Rosie Maternity Hosptial, Addenbrookes, Cambridge
  - University Hospital Coventry, Coventry
  - Darent Valley Hospital, Dartford
  - Simpson Centre for Reproductive Health NHS Lothian, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Medway Maritime Hospital, Gillingham
  - Princess Royal Hospital, Haywards Heath
  - Leeds centre for Newborn Care (Leeds General Infirmary), Leeds
  - Leicester Royal Infirmary, Leicester
  - Liverpool Women's Hospital, Liverpool
  - Homerton University Hospital, London
  - Imperial College Healthcare NHS FT, London
  - Newham General Hosptial, London
  - Northwick Park Hospital, London
  - Queen's Hospital, Barking, London
  - Royal London Hospital, London
  - St Thomas Hospital, London
  - Whipps Cross Hospital, London
  - Luton and Dunstable Hospital, Luton
  - St Mary's Hospital, Manchester
  - Wythenshawe Hosptial, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queens Medical Centre Nottingham, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hosptial, Plymouth
  - Turnbridge Wells Hospital, Royal Tunbridge Wells
  - University Hospital of Wales, Wales
  - Whiston Hospital, Whiston
  - Royal Albert Edward Infirmary, Wigan
  - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Montaldo P, Cirillo M, Burgod C, Caredda E, Ascione S, Carpentieri M, Puzone S, D'Amico A, Garegrat R, Lanza M, Moreno Morales M, Atreja G, Shivamurthappa V, Kariholu U, Aladangady N, Fleming P, Mathews A, Palanisami B, Windrow J, Harvey K, Soe A, Pattnayak S, Sashikumar P, Harigopal S, Pressler R, Wilson M, De Vita E, Shankaran S, Thayyil S; COMET Trial Group. Whole-Body Hypothermia vs Targeted Normothermia for Neonates With Mild Encephalopathy: A Multicenter Pilot Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e249119. doi: 10.1001/jamanetworkopen.2024.9119. PMID 38709535
- [Derived] Garegrat R, Montaldo P, Burgod C, Pant S, Mazlan M, Palanisami B, Chakkarapani E, Woolfall K, Johnson S, Grant PE, Land S, Mahmoud M, Brady T, Cornelius V, Adams E, Dorling J, Aladangadi N, Fleming P, Pressler R, Shennan A, Petrou S, Soe A, Basset P, Shankaran S, Thayyil S. Whole-body hypothermia in mild neonatal encephalopathy: protocol for a multicentre phase III randomised controlled trial. BMC Pediatr. 2024 Jul 18;24(1):460. doi: 10.1186/s12887-024-04935-4. PMID 39026197